CLINICAL TRIAL: NCT00824109
Title: Multicenter Clinical Study Assessing the Performance and the Safety of the Second Generation Antimicrobial Graft in the Abdominal Position
Brief Title: Prospective, Multicenter Study of the Second Generation Antimicrobial Graft in the Abdominal Position
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Datascope Corp. (Industry)
Responsible Party: Philippe Bensimon, Director, Regulatory and Clinical Affairs, and Quality Assurance, Datascope InterVascular
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR07-001
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Aneurysmal Disease of the Abdominal Aorta; Occlusive Disease of the Abdominal Aorta
Keywords: Aneurysmal disease of the abdominal aorta; Occlusive disease of the abdominal aorta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm Study (Other): Consecutive patients meeting the selection criteria
  Interventions: Device: Second Generation Anti-Microbial bifurcated vascular graft (InterGard)

INTERVENTIONS:
Device: Second Generation Anti-Microbial bifurcated vascular graft (InterGard) — treatment of patients with aorto-iliac occlusion,stenosis, or aneurysm
  Other Names: InterGard

SUMMARY:
The purpose of this prospective trial is to demonstrate the safety and performance of the Second Generation Anti-Microbial vascular graft in the treatment of aneurysmal and occlusive diseases of the abdominal aorta.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 - 85 years of age
* Is presenting with an aorto-iliac occlusion (obstruction of flow) or stenosis, or aorto-iliac aneurysm and is eligible for a revascularization with a bifurcated graft
* Is affiliated with a social welfare organization system
* Is willing to participate in the clinical evaluation after signature of the informed consent
* Is able to attend all follow up visits and diagnostics and laboratory exams required by the present protocol

Exclusion Criteria:

* Is treated as an emergency
* Is included in another investigation
* Is pregnant or lactating, or a woman of childbearing potential unwillint to use an effective form of contraception for the duration of the trial
* Has a known allergy to the material device used
* Has previous aorto-iliac bypass or replacement

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Graft patency at three years | three years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Ricco, MD, Principal Investigator — Vascular Surgery Dept, CHU La Miletrie
Locations (1):
- CHU La Miletrie, 350 av. Jacques Coeur, 86021 Poitiers, France